CLINICAL TRIAL: NCT03834636
Title: Impact of Patients Risk Factors, Type of Dental Material and Dental Technique on the Longevity of Aesthetic Dental Restorations
Brief Title: Impact of Patients Risk Factors on the Longevity of Aesthetic Restorations
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, Associate Professor, Principal Investigator, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPGO 029
Record Dates: First submitted 2019-02-07; First posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Dental Restorations Longevity; Dental Restoration Failure; Esthetics, Dental

STUDY DESIGN:
Intervention Model Description: This study is a prospective randomized clinical trial, triple-blind, (patients, investigator and clinical evaluator) with parallel groups. After completing the ICDAS (International Caries Detection and Assessment), clinical occlusal stress examination and questionnaire application on occlusal stress, patients will be randomly divided into two types of dental adhesives and two types of composite resin. Randomization will be stratified according to the risk of caries determined by the ICDAS and the type of cavity to be filled. Operators (Master students and undergraduate students from the last year of the School of Dentistry, Federal University of Pelotas) will place the restorations supervised by highly trained clinicians.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nanoparticulated composite - self-etch (Active Comparator)
  Interventions: Procedure: Restorations with nanoparticulated composites and self etch adhesives
- Nanoparticulated composite - total-etch (Active Comparator)
  Interventions: Procedure: Restorations with nanoparticulated composites and total-etch adhesives
- Nanohybrid composite - self-etch (Active Comparator)
  Interventions: Procedure: Restorations with nanohybrid composites and self etch adhesives
- Nanohybrid composite - total-etch (Active Comparator)
  Interventions: Procedure: Restorations with nanohybrid composites and total-etch adhesives

INTERVENTIONS:
Procedure: Restorations with nanoparticulated composites and self etch adhesives — The restorations will be placed according to the protocol developed for the care, following the guidelines of the manufacturers, with a self-etching dental adhesive (SingleBond Universal, 3M ESPE), selective enamel etching, and use of a nanoparticulated composite (Z350, 3M ESPE)
  Arms: Nanoparticulated composite - self-etch
Procedure: Restorations with nanoparticulated composites and total-etch adhesives — The restorations will be placed according to the protocol developed for the care, following the guidelines of the manufacturers, with a total-etching dental adhesive (SingleBond 2, 3M ESPE), and use of a nanoparticulated composite (Z350, 3M ESPE)
  Arms: Nanoparticulated composite - total-etch
Procedure: Restorations with nanohybrid composites and self etch adhesives — The restorations will be placed according to the protocol developed for the care, following the guidelines of the manufacturers, with a self-etching dental adhesive (SingleBond Universal, 3M ESPE), selective enamel etching, and use of a nanohybrid composite (IPS Empress Direct, Ivoclar Vivadent).
  Arms: Nanohybrid composite - self-etch
Procedure: Restorations with nanohybrid composites and total-etch adhesives — The restorations will be placed according to the protocol developed for the care, following the guidelines of the manufacturers, with a total-etching dental adhesive (SingleBond 2, 3M ESPE), and use of a nanohybrid composite (IPS Empress Direct, Ivoclar Vivadent).
  Arms: Nanohybrid composite - total-etch

SUMMARY:
The objective of this double-blind randomized clinical trial is to evaluate the influence of caries risk, occlusal stress and missing teeth on anterior restorations over a 10 years follow up period. 300 teeth will be randomized according to two adhesive systems: Single Bond 2 and Single Bond Universal (3M ESPE); and two composite resins: nanoparticulated (Filtek ™ Z-350- 3M ESPE) and nanohybrid (IPS Empress Direct - Ivoclar Vivadent). The randomization will be stratified according to the risk of caries and cavity type. The primary outcomes will be longevity, annual failure rate (AFR) and the success of the restorations, and the secondary outcome will be causes for restorations' failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with restorative needs in anterior teeth;
* Patients able to understand and sign the informed consent form;
* Patients willing to return to follow up.

Exclusion Criteria:

* Patients who had a need for Class III and Class IV restorations that did not involve at least 1/3 of the tooth;
* Patients under orthodontic treatment;
* Patients with a compromised general health condition, presenting a greater risk than ASA II, according to the ASA-PS (American Society of Anesthesiologists - Physical Status);
* Patients who had no occlusal contact with an opposing tooth and/or crown;
* Patient with absence of bilateral balanced occlusion;
* Patient with deep caries lesions in close contact with the dental pulp and in need of expectant treatment or direct pulp capping;
* Patients with post-retained need in anterior teeth.

Ages: 9 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-01-10 (Actual); Primary Completion 2022-01-10 (Estimated); Study Completion 2022-01-10 (Estimated)

PRIMARY OUTCOMES:
Survival of the restorations | Changes in the dental restorations status compared to baseline will be assessed yearly up to 10 years.
  Survival of the restoration is defined as any case where the restoration remains functional in the mouth at the time of evaluation, regardless of need of small interventions, such as repair or refurbishment. The restorations were evaluated shortly after baseline and in prospective periods through a direct clinical inspection, with an explorer probe and a clinical mirror, according to the criteria for clinical evaluation of restorations proposed by the FDI (International Dental Federation) (Hickel et al., 2010), the risks of caries and occlusal stress were also evaluated again.
  Two trained and calibrated evaluators, unrelated to making the restorations, blinded to the type of material used, independently performed the clinical evaluations.
Success of the restorations | Changes in the dental restorations status compared to baseline will be assessed yearly up to 10 years.
  Success of the restoration is defined as any case where the restoration remains functional in the mouth at the time of evaluation, without any need of new interventions, and attending the patients demands. The restorations were evaluated shortly after baseline and in prospective periods through a direct clinical inspection, with an explorer probe and a clinical mirror, according to the criteria for clinical evaluation of restorations proposed by the FDI (International Dental Federation) (Hickel et al., 2010), the risks of caries and occlusal stress were also evaluated again.

SECONDARY OUTCOMES:
Patient satisfaction with the treatment | Changes in the patient's satisfaction status compared to baseline will be assessed yearly up to 10 years.
  Patient satisfaction will be recorded with FDI criteria

CONTACTS AND LOCATIONS:
Overall Officials: Maximiliano S Cenci, Principal Investigator — Graduate Program in Dentistry - Federal University of Pelotas
Locations (1):
- Federal Univeristy of Pelotas, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided